CLINICAL TRIAL: NCT05445440
Title: A Phase 1, Two-part, Open-label, Drug-drug Interaction Study in Healthy Male Adult Participants to Evaluate the Effects of BMS-986371 on the Pharmacokinetics of Methotrexate in the Presence and Absence of Sulfasalazine
Brief Title: A Study to Assess the Effects of BMS-986371 on the Drug Levels of Methotrexate in the Presence and Absence of Sulfasalazine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM046-003
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Methotrexate; Leucovorin; Sulfasalazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental)
  Interventions: Drug: Methotrexate; Drug: Leucovorin; Drug: BMS-986371
- Part 2 (Experimental)
  Interventions: Drug: Methotrexate; Drug: Leucovorin; Drug: BMS-986371; Drug: Sulfasalazine

INTERVENTIONS:
Drug: Methotrexate — Specified dose on specified days
Drug: Leucovorin — Specified dose on specified days
Drug: BMS-986371 — Specified dose on specified days
  Other Names: CC-99677
Drug: Sulfasalazine — Specified dose on specified days
  Arms: Part 2

SUMMARY:
The purpose of this study is to evaluate the effects of BMS-986371 on the drug levels of methotrexate, sulfasalazine and their main metabolites in healthy male adult participants.

DETAILED DESCRIPTION:
This study will allow investigation of potential drug-drug interaction mediated through drug transporter proteins. During each part, blood samples will be collected at prespecified times for pharmacokinetic assessments. Subject safety will be monitored throughout the study. There will be approximately 16 subjects enrolled into each part.

ELIGIBILITY:
Inclusion Criteria:

* Participant has physical exam, vital signs, clinical laboratory safety and other medical test results that are within normal limits, considered not clinically significant by the Investigator, or within other parameters specified in the protocol
* Body mass index of 18 to 32 kg/m^2, inclusive

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Current or recent (within 3 months of study intervention administration) gastrointestinal disease that could possibly affect the absorption, distribution, metabolism and excretion of study drug
* Any other medical, psychiatric and/or social reason as determined by the Investigator

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC[0-T]) | Up to 22 days
  Part 1
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC[INF]) | Up to 22 days
  Part 1
Maximum observed plasma concentration (Cmax) | Up to 22 days
  Part 1

SECONDARY OUTCOMES:
AUC(0-T) | Up to 22 days
  Part 2
AUC(INF) | Up to 22 days
  Part 2
Cmax | Up to 22 days
  Part 2
Number of participants with adverse events (AEs) | Up to 30 days post participant's last study treatment
  Parts 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Quotient Sciences Miami, Miami, Florida, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/us/en/home.html